CLINICAL TRIAL: NCT00705965
Title: A Stepwise Psychotherapy Intervention for Reducing Risk in Coronary Artery Disease - a Randomised Controlled Trial (SPIRR-CAD)
Brief Title: Effects of a Psychotherapy Intervention in Depressed Patients With Coronary Artery Disease
Acronym: SPIRR-CAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Göttingen (Other)
Collaborators: University of Cologne (Other); Johannes Gutenberg University Mainz (Other); Humboldt-Universität zu Berlin (Other); University Hospital Freiburg (Other); Kerckhoff Rehabilitation Center Bad Nauheim (Unknown); Heidelberg University (Other); Hannover Medical School (Other); Technical University of Munich (Other); Technische Universität Dresden (Other); Nuremberg General Hospital (Unknown); The Clinical Trials Centre Cologne (Other); German Research Foundation (Other); Medical University of Graz (Other)
Responsible Party: Principal Investigator, Christoph Herrmann-Lingen, Professor Dr., University of Göttingen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZKSK-371
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Depression; Coronary Artery Disease
Keywords: Coronary artery disease; depression; psychotherapy; randomized controlled trial
MeSH Terms: conditions — Depression; Coronary Artery Disease | interventions — Psychotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Stepwise, manualized individual and group psychotherapy in addition to usual cardiological care.
  Interventions: Behavioral: Psychotherapy; Other: Usual cardiological care
- 2 (Active Comparator): Usual cardiological care including one information session.
  Interventions: Behavioral: Information session; Other: Usual cardiological care

INTERVENTIONS:
Behavioral: Psychotherapy — Stepwise, manualized individual and group psychotherapy in addition to usual cardiological care.
  Other Names: Stepwise manualized psychotherapy
  Arms: 1
Behavioral: Information session — One information session about living with heart disease.
  Arms: 2
Other: Usual cardiological care — Usual cardiological care

SUMMARY:
In patients with coronary artery disease (CAD), depressive symptoms are frequent and highly relevant for quality of life, health behaviour, health care costs, and prognosis. The aim of the current study is to evaluate the effects of a psychotherapy intervention on symptoms of depression in patients with CAD. Therefore, depressed patients diagnosed with CAD will be randomised into a controlled intervention trial, comparing a stepwise psychotherapy intervention with usual cardiological care. The manualized psychotherapy intervention starts with three individual sessions offered on a weekly basis. Afterwards, symptoms of depression will be re-evaluated and, in case of persisting symptoms, patients receive an additional 25 sessions of psychodynamic group psychotherapy over a total period of one year. The psychodynamic approach was chosen in order to specifically take into account personality traits such as negative affectivity and social inhibition, the components of the Type D personality, which may explain why recent cognitive behavioural psychotherapy (CBT) trials produced only small effects in depressed CAD patients. The investigators expect that the intervention will reduce depressive symptoms as well as the prevalence of depressive disorders. It will also improve both behaviourally and physiologically mediated cardiovascular risk indicators, promote better quality of life, and reduce healthcare costs. Subgroup analyses will be performed in order to identify gender-specific treatment effects, effects on immunological stress reactivity, and genetic predictors of treatment success.

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary artery disease
* German speaking men and women
* Recent coronary angiogram (<= 3 months old)
* Depression score (HADS-D) >= 8
* Written informed consent

Exclusion Criteria:

* Severe heart failure
* Other acutely life- threatening conditions
* Severe chronic inflammatory disease
* Current suicidal tendency
* Severe depressive episode
* Other severe mental illness.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Actual)
Dates: Start 2008-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Changes from baseline to 18 months in depressive symptoms (HADS-D) | 18 months

SECONDARY OUTCOMES:
Remission of depressive disorder (SCID) and the Type D pattern (DS-14), reduced severity of depressive symptoms (HAM-D) | 18 months
Health-related quality of life (SF36, EuroQuol-5D) | 18 months
cardiovascular risk profile | 18 months
neuroendocrine and immunological activation | 18 months
coagulation | 18 months
heart rate variability | 18 months
cardiac events | 18 months
health care utilisation and costs | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Herrmann-Lingen, MD, Principal Investigator — University of Goettingen, Dept. of Psychosomatic Medicine and Psychotherapy; Christian Albus, MD, Principal Investigator — University of Cologne, Dept. of Psychosomatics and Psychotherapy
Locations (10):
- Germany (10):
  - Berlin University Medical Center, Campus Benjamin Franklin, Dept. of Psychosomatics and Psychotherapy, Berlin
  - University of Cologne, Dept. Psychosomatics and Psychotherapy, Cologne
  - Technical University of Dresden, Dept. of Psychotherapy and Psychosomatics, Dresden
  - University Hospital of Freiburg, Dept. of Psychosomatic Medicine and Psychotherapy, Freiburg im Breisgau
  - University of Goettingen, Dept. of Psychosomatic Medicine and Psychotherapy, Göttingen
  - Hannover Medical School, Dept. of Psychosomatics and Psychotherapy, Hanover
  - University of Heidelberg, Dept. of General Internal and Psychosomatic Medicine, Heidelberg
  - University Hospital of Mainz, Dept. of Psychosomatic Medicine and Psychotherapy, Mainz
  - Technical University of Munich, Institute and Dept. of Psychosomatic Medicine, Psychotherapy and Medical Psychology, München
  - Nuremberg General Hospital, Department of Psychosomatic Medicine and Psychotherapy, Nuremberg

REFERENCES:
- [Background] Albus C, Beutel ME, Deter HC, Fritzsche K, Hellmich M, Jordan J, Juenger J, Krauth C, Ladwig KH, Michal M, Mueck-Weymann M, Petrowski K, Pieske B, Ronel J, Soellner W, Waller C, Weber C, Herrmann-Lingen C. A stepwise psychotherapy intervention for reducing risk in coronary artery disease (SPIRR-CAD) - rationale and design of a multicenter, randomized trial in depressed patients with CAD. J Psychosom Res. 2011 Oct;71(4):215-22. doi: 10.1016/j.jpsychores.2011.02.013. Epub 2011 Apr 15. PMID 21911098
- [Result] Herrmann-Lingen C, Beutel ME, Bosbach A, Deter HC, Fritzsche K, Hellmich M, Jordan J, Junger J, Ladwig KH, Michal M, Petrowski K, Pieske B, Ronel J, Sollner W, Stohr A, Weber C, de Zwaan M, Albus C; SPIRR-CAD Study Group. A Stepwise Psychotherapy Intervention for Reducing Risk in Coronary Artery Disease (SPIRR-CAD): Results of an Observer-Blinded, Multicenter, Randomized Trial in Depressed Patients With Coronary Artery Disease. Psychosom Med. 2016 Jul-Aug;78(6):704-15. doi: 10.1097/PSY.0000000000000332. PMID 27187851
- [Derived] Fangauf SV, Meyer T, Albus C, Binder L, Deter HC, Ladwig KH, Michal M, Ronel J, Rothenberger A, Sollner W, Wachter R, Weber CS, Herrmann-Lingen C; SPIRR-CAD group. Longitudinal relationship between B-type natriuretic peptide and anxiety in coronary heart disease patients with depression. J Psychosom Res. 2019 Aug;123:109728. doi: 10.1016/j.jpsychores.2019.05.006. Epub 2019 May 21. PMID 31376874
- [Derived] Vitinius F, Escherich S, Deter HC, Hellmich M, Junger J, Petrowski K, Ladwig KH, Lambertus F, Michal M, Weber C, de Zwaan M, Herrmann-Lingen C, Ronel J, Albus C. Somatic and sociodemographic predictors of depression outcome among depressed patients with coronary artery disease - a secondary analysis of the SPIRR-CAD study. BMC Psychiatry. 2019 Feb 4;19(1):57. doi: 10.1186/s12888-019-2026-6. PMID 30717711
- [Derived] Sollner W, Muller MM, Albus C, Behnisch R, Beutel ME, de Zwaan M, Fritzsche K, Habermeier A, Hellmich M, Jordan J, Junger J, Ladwig KH, Michal M, Petrowski K, Ronel J, Stein B, Weber C, Weber R, Herrmann-Lingen C. The relationship between attachment orientations and the course of depression in coronary artery disease patients: A secondary analysis of the SPIRR-CAD trial. J Psychosom Res. 2018 May;108:39-46. doi: 10.1016/j.jpsychores.2018.02.014. Epub 2018 Feb 24. PMID 29602324
- [Derived] Orth-Gomer K, Deter HC, Grun AS, Herrmann-Lingen C, Albus C, Bosbach A, Ladwig KH, Ronel J, Sollner W, de Zwaan M, Petrowski K, Weber C; SPIRR-CAD Study Group. Socioeconomic factors in coronary artery disease - Results from the SPIRR-CAD study. J Psychosom Res. 2018 Feb;105:125-131. doi: 10.1016/j.jpsychores.2017.12.005. Epub 2017 Dec 5. PMID 29332628
- [Derived] Lambertus F, Herrmann-Lingen C, Fritzsche K, Hamacher S, Hellmich M, Junger J, Ladwig KH, Michal M, Ronel J, Schultz JH, Vitinius F, Weber C, Albus C. Prevalence of mental disorders among depressed coronary patients with and without Type D personality. Results of the multi-center SPIRR-CAD trial. Gen Hosp Psychiatry. 2018 Jan-Feb;50:69-75. doi: 10.1016/j.genhosppsych.2017.10.001. Epub 2017 Oct 7. PMID 29078170
- Available data/document: treatment manual and supplemental content — http://links.lww.com/PSYMED/A275